CLINICAL TRIAL: NCT00464269
Title: An International, Double-blind, Parallel-group, Placebo-controlled, Randomized Study: Evaluation of the Efficacy and Safety of Brivaracetam in Subjects (>= 16 to 70 Years Old) With Partial Onset Seizures
Brief Title: Double-blind, Randomized Study Evaluating the Efficacy and Safety of Brivaracetam in Adults With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01253; 2006-006345-14 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Partial Onset Seizures, Adolescents & Adults
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Matching Placebo tablets administered twice a day. Daily oral dose of two equal intakes, morning and evening, of Placebo in a double-blinded way for the 12-week Treatment Period.
  Interventions: Other: Placebo
- Brivaracetam 5 mg/day (Experimental): Brivaracetam 5 mg/day, 2.5 mg administered twice a day. Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 5 mg /day in a double-blinded way for the 12-week Treatment Period.
  Interventions: Drug: Brivaracetam 2.5 mg
- BRV 20mg/day (Experimental): Brivaracetam 20 mg/day, 10 mg administered twice a day. Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 20 mg /day in a double-blinded way for the 12-week Treatment Period.
  Interventions: Drug: Brivaracetam 10 mg
- BRV 50mg/day (Experimental): Brivaracetam 50 mg/day, 25 mg administered twice a day. Daily oral dose of two equal intakes, morning and evening, of Brivaracetam 50 mg /day, in a double-blinded way for the 12-week Treatment Period.
  Interventions: Drug: Brivaracetam 25 mg

INTERVENTIONS:
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 2.5 mg, 10 mg and 25 mg
  * Route of Administration: Oral use
  Arms: Placebo
Drug: Brivaracetam 2.5 mg — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 2.5 mg
  * Route of Administration: Oral use
  Arms: Brivaracetam 5 mg/day
Drug: Brivaracetam 10 mg — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 10 mg
  * Route of Administration: Oral use
  Arms: BRV 20mg/day
Drug: Brivaracetam 25 mg — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 25 mg
  * Route of Administration: Oral use
  Arms: BRV 50mg/day

SUMMARY:
This study will evaluate the efficacy and safety of Brivaracetam to support the submission file in the indication of adjunctive treatment in adolescents and adults with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were 16 to 70 years, both inclusive. Subjects under 18 years of age were only included where legally permitted and ethically accepted
* Subjects with well-characterized focal epilepsy or epileptic syndrome according to the International League Against Epilepsy (ILAE) classification
* Subjects had a history of partial onset seizures (POS) whether or not secondarily generalized (Type I seizures according to the ILAE classification)
* Subjects had at least 2 POS whether or not secondarily generalized per month during the 3 months preceding Visit 1 (V1)
* Subjects had at least 8 POS whether or not secondarily generalized during the 8-Week Baseline Period
* Subjects were uncontrolled while treated by 1 to 2 permitted concomitant antiepileptic drug(s) (AEDs). Vagal nerve stimulation (VNS) was allowed and was not counted as a concomitant AED

Exclusion Criteria:

* History or presence of seizures occurring only in clusters (too frequently or indistinctly separated to be reliably counted) before Visit 3
* History or presence of status epilepticus during the year preceding Visit 1 or during Baseline

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (69):
- United States (40):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - Los Angeles, California
  - Newport Beach, California
  - Sacramento, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Saint Paul, Minnesota
  - Tupelo, Mississippi
  - Chesterfield, Missouri
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (9):
  - Chatswood, New South Wales
  - Randwick, New South Wales
  - Woodville, South Australia
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Parkville, Victoria
  - Adelaide
  - Fitzroy
  - West Heidelberg
- Brazil (8):
  - Campinas
  - Curitiba
  - Florianópolis
  - Porto Alegre
  - Ribeirão Preto
  - Salvador
  - São José do Rio Preto
  - São Paulo
- Canada (4):
  - Edmonton, Alberta
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
- Mexico (8):
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Aguascalientes
  - Chihuahua City
  - Mexico City
  - Monterrey
  - Nuevo León
  - San Luis Potosí City

REFERENCES:
- [Result] Biton V, Berkovic SF, Abou-Khalil B, Sperling MR, Johnson ME, Lu S. Brivaracetam as adjunctive treatment for uncontrolled partial epilepsy in adults: a phase III randomized, double-blind, placebo-controlled trial. Epilepsia. 2014 Jan;55(1):57-66. doi: 10.1111/epi.12433. Epub 2013 Nov 8. PMID 24446953
- [Result] Toledo M, Whitesides J, Schiemann J, Johnson ME, Eckhardt K, McDonough B, Borghs S, Kwan P. Safety, tolerability, and seizure control during long-term treatment with adjunctive brivaracetam for partial-onset seizures. Epilepsia. 2016 Jul;57(7):1139-51. doi: 10.1111/epi.13416. Epub 2016 Jun 6. PMID 27265725
- [Result] Ben-Menachem E, Mameniskiene R, Quarato PP, Klein P, Gamage J, Schiemann J, Johnson ME, Whitesides J, McDonough B, Eckhardt K. Efficacy and safety of brivaracetam for partial-onset seizures in 3 pooled clinical studies. Neurology. 2016 Jul 19;87(3):314-23. doi: 10.1212/WNL.0000000000002864. Epub 2016 Jun 22. PMID 27335114
- [Result] Brodie MJ, Whitesides J, Schiemann J, D'Souza J, Johnson ME. Tolerability, safety, and efficacy of adjunctive brivaracetam for focal seizures in older patients: A pooled analysis from three phase III studies. Epilepsy Res. 2016 Nov;127:114-118. doi: 10.1016/j.eplepsyres.2016.08.018. Epub 2016 Aug 18. PMID 27589414
- [Result] Mukuria C, Young T, Keetharuth A, Borghs S, Brazier J. Sensitivity and responsiveness of the EQ-5D-3L in patients with uncontrolled focal seizures: an analysis of Phase III trials of adjunctive brivaracetam. Qual Life Res. 2017 Mar;26(3):749-759. doi: 10.1007/s11136-016-1483-3. Epub 2016 Dec 21. PMID 28004320
- [Result] Moseley BD, Sperling MR, Asadi-Pooya AA, Diaz A, Elmouft S, Schiemann J, Whitesides J. Efficacy, safety, and tolerability of adjunctive brivaracetam for secondarily generalized tonic-clonic seizures: Pooled results from three Phase III studies. Epilepsy Res. 2016 Nov;127:179-185. doi: 10.1016/j.eplepsyres.2016.09.003. Epub 2016 Sep 3. PMID 27608437
- [Result] Brandt C, Borghs S, Elmoufti S, Mueller K, Townsend R, de la Loge C. Health-related quality of life in double-blind Phase III studies of brivaracetam as adjunctive therapy of focal seizures: A pooled, post-hoc analysis. Epilepsy Behav. 2017 Apr;69:80-85. doi: 10.1016/j.yebeh.2016.11.031. Epub 2017 Feb 23. PMID 28236727
- [Result] Klein P, Johnson ME, Schiemann J, Whitesides J. Time to onset of sustained >/=50% responder status in patients with focal (partial-onset) seizures in three phase III studies of adjunctive brivaracetam treatment. Epilepsia. 2017 Feb;58(2):e21-e25. doi: 10.1111/epi.13631. Epub 2016 Dec 18. PMID 27988967
- [Result] Asadi-Pooya AA, Sperling MR, Chung S, Klein P, Diaz A, Elmoufti S, Schiemann J, Whitesides J. Efficacy and tolerability of adjunctive brivaracetam in patients with prior antiepileptic drug exposure: A post-hoc study. Epilepsy Res. 2017 Mar;131:70-75. doi: 10.1016/j.eplepsyres.2017.02.007. Epub 2017 Feb 27. PMID 28279891
- [Result] Benbadis S, Klein P, Schiemann J, Diaz A, Elmoufti S, Whitesides J. Efficacy, safety, and tolerability of brivaracetam with concomitant lamotrigine or concomitant topiramate in pooled Phase III randomized, double-blind trials: A post-hoc analysis. Epilepsy Behav. 2018 Mar;80:129-134. doi: 10.1016/j.yebeh.2017.12.024. Epub 2018 Feb 3. PMID 29414542
- [Result] Brodie MJ, Fakhoury T, McDonough B, Colson AO, Stockis A, Elmoufti S, Whitesides J. Brivaracetam-induced elevation of carbamazepine epoxide levels: A post-hoc analysis from the clinical development program. Epilepsy Res. 2018 Sep;145:55-62. doi: 10.1016/j.eplepsyres.2018.06.002. Epub 2018 Jun 4. PMID 29908435
- [Result] Klein P, Laloyaux C, Elmoufti S, Gasalla T, Martin MS. Time course of 75%-100% efficacy response of adjunctive brivaracetam. Acta Neurol Scand. 2020 Aug;142(2):175-180. doi: 10.1111/ane.13287. Epub 2020 Jun 9. PMID 32432339
- [Result] Moseley BD, Dimova S, Elmoufti S, Laloyaux C, Asadi-Pooya AA. Long-term efficacy and tolerability of adjunctive brivaracetam in adults with focal to bilateral tonic-clonic (secondary generalized) seizures: Post hoc pooled analysis. Epilepsy Res. 2021 Oct;176:106694. doi: 10.1016/j.eplepsyres.2021.106694. Epub 2021 Jun 24. PMID 34218211
- [Result] Ryvlin P, Dimova S, Elmoufti S, Floricel F, Laloyaux C, Nondonfaz X, Biton V. Tolerability and efficacy of adjunctive brivaracetam in adults with focal seizures by concomitant antiseizure medication use: Pooled results from three phase 3 trials. Epilepsia. 2022 Aug;63(8):2024-2036. doi: 10.1111/epi.17304. Epub 2022 Jun 10. PMID 35582748
- [Derived] Bresnahan R, Panebianco M, Marson AG. Brivaracetam add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2022 Mar 14;3(3):CD011501. doi: 10.1002/14651858.CD011501.pub3. PMID 35285519
- [Derived] Lee SK, Heo K, Kim SE, Lee SA, Elmoufti S, Laloyaux C, Hur B. Effect of Number of Previous Antiseizure Medications on Efficacy and Tolerability of Adjunctive Brivaracetam for Uncontrolled Focal Seizures: Post Hoc Analysis. Adv Ther. 2021 Jul;38(7):4082-4099. doi: 10.1007/s12325-021-01816-5. Epub 2021 Jun 21. PMID 34155568
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in September 2007 and concluded in January 2009. 400 subjects were randomized of which 396 are included in the Safety Population.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS).
Groups:
- Placebo: Matching Placebo tablets administered twice a day
- BRV 5 mg/Day: Brivaracetam 5 mg/day, 2.5 mg administered twice a day
- BRV 20 mg/Day: Brivaracetam 20 mg/day, 10 mg administered twice a day
- BRV 50 mg/Day: Brivaracetam 50 mg/day, 25 mg administered twice a day
Period: Overall Study
Arm/Group | Placebo | BRV 5 mg/Day | BRV 20 mg/Day | BRV 50 mg/Day
Started | 99 | 99 | 100 | 102
Completed | 93 | 82 | 93 | 93
Not Completed | 6 | 17 | 7 | 9
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Other reason | 3 | 3 | 1 | 1
Not completed — AE, serious fatal | 0 | 0 | 1 | 1
Not completed — SAE, non-fatal | 0 | 0 | 0 | 1
Not completed — AE, non-serious non-fatal | 2 | 8 | 3 | 4
Not completed — SAE,non-fatal+AE,non-serious non-fatal | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Randomized Set.
Arm/Group | Placebo | BRV 5 mg/Day | BRV 20 mg/Day | BRV 50 mg/Day | Total Title
Number analyzed (Participants) | 99 | 99 | 100 | 102 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (12.6) | 38.8 (11.6) | 37.3 (13.3) | 39.0 (12.3) | 38.2 (12.5)
Age, Customized [Number; unit: participants]
  < 18 years | 7 | 0 | 5 | 2 | 14
  18 - < 65 years | 91 | 97 | 93 | 99 | 380
  65 - < 85 years | 1 | 2 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 48 | 50 | 202
  Male | 44 | 50 | 52 | 52 | 198

OUTCOME MEASURES:

1. Primary Outcome: Partial Onset Seizure (Type I) Frequency Per Week Over the 12-week Treatment Period
Description: Partial (Type I) seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to generalized tonic-clonic convulsions.
  Partial Onset Seizure (POS) Frequency per week over the Treatment Period (TP) was calculated as:
  (Total Type I seizures over the TP)*7/(Total number of days with no missing seizure count in the TP)
Time Frame: Baseline to 12-week Treatment Period
Population: The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant GCP deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Groups:
- Modified Intention-to-Treat (Placebo Treated Subjects): Matching Placebo tablets administered twice a day.
  The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant Good Clinical Practice (GCP) deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
- Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects): Brivaracetam (BRV) 5 mg/day, 2.5 mg administered twice a day.
  The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant GCP deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
- Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects): Brivaracetam 20 mg/day, 10 mg administered twice a day.
  The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant GCP deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
- Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects): Brivaracetam 50 mg/day, 25 mg administered twice a day.
  The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant GCP deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
seizures per week | 2.15 [1.43 to 4.15] | 1.80 [0.99 to 5.59] | 1.96 [1.05 to 5.45] | 1.70 [0.91 to 4.80]
Statistical Analysis 1: Comparison: Modified Intention-to-Treat (Placebo Treated Subjects) vs Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects); The treatment difference between each Brivaracetam (BRV) dose and Placebo (PBO) is reported as a percent reduction over Placebo. The treatment effect was estimated using the 95 % confidence intervals; Test type: Non-Inferiority or Equivalence — The overall significance level was controlled at 5 %. The 3 doses of Brivaracetam were tested at the 5 % level against Placebo starting from the 50 mg dose then the 20 mg dose and finally the 5 mg dose, only moving to the next test if the previous one is significant at the 5 % level; p = 0.025, ANCOVA; Baseline and Treatment Period Partial Onset Seizure (POS) frequencies are standardized to a 7-day duration; % reduction over Placebo = 12.8, 95% CI 2-sided [1.7 to 22.6] — The log-transformed (log(x+1)) POS seizure frequency was analyzed using an ANCOVA model, including terms for treatment, stratification factors, and log-transformed Baseline POS seizure frequency per week as a covariate
Statistical Analysis 2: Comparison: Modified Intention-to-Treat (Placebo Treated Subjects) vs Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects); The treatment difference between each Brivaracetam dose an Placebo is reported as a percent reduction over Placebo. The treatment effect was estimated using 95 % confidence intervals; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.492, ANCOVA; Baseline and Treatment Period Partial Onset Seizure (POS) frequencies are standardized to 7-day duration; % reduction over Placebo = 4.1, 95% CI 2-sided [-8.1 to 15.0] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Responder Rate for Partial Onset Seizure (Type I) Frequency Per Week Over the 12-week Treatment Period
Description: The responder rate was presented as the number of responders and non-responders. A subject is a responder, if the subject has at least 50 % reduction in partial onset seizure frequency per week from Baseline to Treatment Period. Subjects with zero seizure frequency per week at Baseline were considered as non-responders.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Modified Intention-to-Treat (Placebo Treated Subjects): Matching Placebo tablets administered twice a day.
  The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant GCP deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
- Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects): Brivaracetam 5 mg/day, 2.5 mg administered twice a day.
  The modified Intent-To-Treat population consists of subjects who received at least one dose of study medication but excluding 3 randomized subjects from a site with significant GCP deviations and 1 subject who had an exceedingly high seizure frequency and a clinical presentation that may not have been consistent with a diagnosis of focal epilepsy.
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
participants
  Responders | 16 | 21 | 23 | 33
  Non-responders | 80 | 75 | 76 | 68

3. Secondary Outcome: All Seizure Frequency (Type I+II+III) Per Week Over the 12-week Treatment Period
Description: There are three different types of seizures:
  * Type I: Partial seizures
  * Type II: Generalized seizures
  * Type III: Unclassified epileptic seizures.
  All seizure frequency per week over Treatment Period (TP) was calculated as: (Total number of seizures over the TP)*7/(Total number of days with no missing seizure count in the TP)
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
seizures per week | 2.15 [1.45 to 4.23] | 1.80 [0.99 to 5.59] | 1.96 [1.05 to 5.85] | 1.77 [0.99 to 4.80]

4. Secondary Outcome: Percent Change From Baseline to the 12-week Treatment Period in Partial Onset Seizure (Type I) Frequency Per Week
Description: Percent change from Baseline was calculated as percent reduction by:
  (weekly seizure frequency Baseline - weekly seizure frequency Treatment)*100/(weekly seizure frequency Baseline).
  The higher the values for percent change in Partial Onset Seizure (POS) frequency, the higher the improvement from Baseline.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change in POS frequency
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 95 | 96 | 99 | 101
Percent change in POS frequency | 17.75 [-5.11 to 37.07] | 19.95 [-12.96 to 45.15] | 22.52 [-4.56 to 46.51] | 30.47 [11.40 to 59.78]

5. Secondary Outcome: Categorized Percentage Change From Baseline in Seizure Frequency for Partial Onset Seizure (Type I) Over the 12-week Treatment Period
Description: Subjects were classified in 1 of the following categories based on their percent reduction from Baseline to Treatment Period in Partial Onset Seizure (POS) frequency per week: <-25 %, -25 % to <25 %, 25 % to <50 %, 50 % to <75 %, 75 % to <100 %, and 100 %.
  Subjects having zero for Baseline seizure frequency per week were classified in the <-25 % category.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
percentage of participants
  <-25 % | 14.6 | 21.9 | 14.1 | 9.9
  -25 % to < 25 % | 44.8 | 31.3 | 38.4 | 31.7
  25 % to < 50 % | 24.0 | 25.0 | 24.2 | 25.7
  50 % to < 75 % | 12.5 | 12.5 | 15.2 | 19.8
  75 % to < 100 % | 4.2 | 8.3 | 6.1 | 8.9
  100 % | 0 | 1.0 | 2.0 | 4.0

6. Secondary Outcome: Seizure Freedom Rate (All Seizure Types) Over the 12-week Treatment Period
Description: Subjects were considered seizure free if their seizure counts for every day over the Treatment Period (TP) was zero and if they did not discontinue before the end of the TP. Seizure freedom rate was calculated as:
  (total number of seizure - free subjects in treatment group during TP)/(total number of evaluable Intent-To-Treat (ITT) subjects in treatment group)
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
percentage of participants
  Seizure-free | 0 | 1.0 | 1.0 | 4.0
  No seizures but non-completer | 0 | 0 | 1.0 | 0
  Not seizure-free | 100.0 | 99.0 | 98.0 | 96.0

7. Secondary Outcome: Time to First Type I Seizure During the 12-week Treatment Period
Description: The time to first Partial Onset Seizure (POS) in the Treatment Period is defined as the time between beginning of the Treatment Period and the date of occurrence of first Type I seizure. Subjects withdrawing during the Treatment Period before having a first Type I seizure were considered as having a first Type I seizure on the last day of their Treatment Period.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
days | 3 [2 to 3] | 4 [2 to 5] | 5 [3 to 7] | 4 [3 to 6]

8. Secondary Outcome: Time to Fifth Type I Seizure During the 12-week Treatment Period
Description: The time to fifth Partial Onset Seizure (POS) in the Treatment Period is defined as the time between beginning of the Treatment Period and the date of occurrence of fifth Type I seizure. Subjects withdrawing during the Treatment Period before having a fifth Type I seizure were considered as having a fifth Type I seizure on the last day of their Treatment Period.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
days | 15 [12 to 16] | 14 [12 to 18] | 17 [14 to 21] | 19 [16 to 25]

9. Secondary Outcome: Time to Tenth Type I Seizure During the 12-week Treatment Period
Description: The time to tenth Partial Onset Seizure (POS) in the Treatment Period is defined as the time between beginning of the Treatment Period and the date of occurrence of tenth Type I seizure. Subjects withdrawing during the Treatment Period before having a tenth Type I seizure were considered as having a tenth Type I seizure on the last day of their Treatment Period.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 96 | 96 | 99 | 101
days | 28 [24 to 33] | 30 [21 to 38] | 34 [25 to 46] | 37 [27 to 52]

10. Secondary Outcome: Reduction of Type IC/Type I Seizure Frequency Ratio From Baseline to the 12- Week Treatment Period
Description: The type IC/Type I seizure frequency ratio is represented by the percentage of subjects having a reduction in the ratio of Type IC seizure frequency over Type IA, IB, and IC seizure frequency from Baseline to Treatment Period.
Time Frame: Baseline to 12-week Treatment Period
Population: The Intention-to-treat (ITT) population was defined as all randomized subjects who received at least 1 dose of study medication.
  Type IC Population consists of those subjects with at least one Type IC seizure during the Baseline period.
Measure: Number; unit: percentage of participants
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 32 | 34 | 36 | 33
percentage of participants | 56.3 | 50.0 | 77.8 | 63.6

11. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Total Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: The Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) is an adaptation of the original QOLIE-31 instrument that includes 30 items grouped into seven multi-items subscales - seizure worry (5 items), overall quality of life (2 items), emotional well-being (5 items), energy / fatigue (4 items), cognitive functioning (6 items), medication effects (3 items), and social function (5 items) - and a health status item.
  The subscale scores, the total score and the health status item score range from 0 to 100 and higher scores indicating better function.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 86 | 81 | 81 | 85
units on a scale | 3.88 (14.44) | 4.07 (15.40) | 5.19 (15.47) | 2.88 (13.53)

12. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Seizure Worry Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 84 | 84 | 86
units on a scale | 9.36 (26.98) | 3.34 (19.20) | 3.69 (24.55) | 5.97 (21.79)

13. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Daily Activities / Social Functioning Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 11
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 84 | 84 | 87
units on a scale | 1.97 (28.39) | 7.03 (23.47) | 7.73 (26.04) | 2.06 (23.02)

14. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Hospital Anxiety Score
Description: The Hospital Anxiety and Depression Scale (HADS) was used to evaluate anxiety and depression. The HADS was developed as a self administered scale to assess the presence and severity of both anxiety and depression simultaneously. It consists of 14 items that are scored on a 4-point severity scale ranging from 0 to 3. A score per dimension was calculated with each score ranging from 0 to 21 and higher scores indicating higher depression / anxiety. A negative value in change from Baseline shows an improvement in HADS from Baseline.
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 84 | 84 | 86
units on a scale | 7.44 (4.32) | 7.32 (4.03) | 6.55 (3.94) | 7.99 (3.63)

15. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Hospital Depression Score
Description: as for outcome 14
Time Frame: Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 84 | 84 | 86
units on a scale | 5.36 (3.78) | 4.97 (4.00) | 4.82 (3.56) | 5.81 (3.70)

16. Secondary Outcome: Patient's Global Evaluation Scale (P-GES) Evaluated at Last Visit or Early Discontinuation Visit
Description: Patient's Global Evaluation Scale (P-GES) is a global assessment of the disease evolution which was performed using a seven-point scale (1= Marked worsening to 7 = Marked improvement) with the start of the study medication as the reference time point. The subject completed it by answering to the following: 'Overall, has there been a change in your seizures since the start of the study medication?'
Time Frame: Baseline to Last Visit or Early Discontinuation Visit in the 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 84 | 81 | 80 | 86
percentage of participants
  Marked improvement | 15.5 | 19.8 | 18.8 | 26.7
  Moderate improvement | 25.0 | 24.7 | 26.3 | 19.8
  Slight improvement | 23.8 | 18.5 | 21.3 | 22.1
  No change | 28.6 | 23.5 | 27.5 | 23.3
  Slight worsening | 4.8 | 6.2 | 1.3 | 4.7
  Moderate worsening | 1.2 | 7.4 | 3.8 | 1.2
  Marked worsening | 1.2 | 0 | 1.3 | 2.3

17. Secondary Outcome: Investigator's Global Evaluation Scale (I-GES) Evaluated at Last Visit or Early Discontinuation Visit
Description: The Investigator's Global Evaluation Scale (I-GES) is a global assessment of the disease evolution which was performed using a seven-point scale (1 = Marked worsening to 7 = Marked improvement) with the start of the study medication as the reference time point. The investigator completed it by answering to the following: 'Assess the overall change in the severity of patient's illness, compared to start of study medication.'
Time Frame: Baseline to Last Visit or Early Discontinuation Visit in the 12-week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 95 | 90 | 99 | 98
percentage of participants
  Marked improvement | 12.6 | 12.2 | 17.2 | 16.3
  Moderate improvement | 20.0 | 18.9 | 18.2 | 27.6
  Slight improvement | 21.1 | 24.4 | 31.3 | 24.5
  No change | 41.1 | 34.4 | 32.3 | 25.5
  Slight worsening | 3.2 | 2.2 | 1.0 | 2.0
  Moderate worsening | 1.1 | 7.8 | 0 | 3.1
  Marked worsening | 1.1 | 0 | 0 | 1.0

18. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Energy/Fatigue Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: The QOLIE-31-P is an adaptation of the original QOLIE-31 instrument that includes 30 items grouped into seven multi-item subscales - Seizure Worry (5 items), Overall Quality of Life (2 items), Emotional Well-Being (5 items), Energy/Fatigue (4 items), Cognitive Functioning (6 items), Medication Effects (3 items) and Daily Activities/Social Functioning (5 items) - and a Health Status item. The subscale scores, the Total score and the Health Status item score are calculated according to the scoring algorithm defined by the author with scores ranging from 0 to 100 and higher scores indicating better function. A positive value in Change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 86 | 82 | 82 | 86
units on a scale | 6.41 (19.55) | 2.24 (23.10) | 3.94 (15.56) | 0.45 (20.07)

19. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Emotional Well-Being Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 18
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 83 | 81 | 87
units on a scale | 2.14 (18.28) | 1.69 (21.61) | 2.07 (19.10) | 1.97 (17.29)

20. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Cognitive Functioning Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 18
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 83 | 84 | 86
units on a scale | 2.79 (20.34) | 4.26 (21.23) | 6.36 (24.61) | 3.37 (19.16)

21. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Medication Effects Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 18
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 84 | 84 | 86
units on a scale | 1.02 (34.05) | -2.61 (28.08) | 0.73 (25.94) | 6.07 (30.90)

22. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Overall Quality of Life Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 18
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 87 | 84 | 84 | 87
units on a scale | 5.49 (16.25) | 3.39 (19.70) | 3.66 (20.10) | 2.33 (19.14)

23. Secondary Outcome: Change From Baseline to the 12-week Treatment Period in Health Status of Life Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 18
Time Frame: From Baseline to 12-week Treatment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified Intention-to-Treat (Placebo Treated Subjects) | Modified Intention-to-Treat (BRV 5 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 20 mg/Day Treated Subjects) | Modified Intention-to-Treat (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 86 | 84 | 84 | 85
units on a scale | 8.1 (22.0) | 6.9 (23.5) | 7.3 (21.1) | 5.5 (20.9)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 23 weeks from Visit 1 (Week -8) to the Safety Visit (Week 15).
Description: Adverse Events (AEs) refer to the Safety Population including all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Placebo | BRV 5 mg/Day | BRV 20 mg/Day | BRV 50 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/98 | 1/97 | 3/100 | 4/101
Other Adverse Events (participants affected / at risk) | 32/98 | 49/97 | 46/100 | 51/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | BRV 5 mg/Day (N=97) | BRV 20 mg/Day (N=100) | BRV 50 mg/Day (N=101)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration bronchial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | BRV 5 mg/Day (N=97) | BRV 20 mg/Day (N=100) | BRV 50 mg/Day (N=101)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 7 (8) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 4 (4) | 4 (5) | 6 (6)
Fatigue (General disorders) | 2 (2) | 3 (3) | 13 (14) | 10 (12)
Influenza (Infections and infestations) | 1 (1) | 9 (10) | 6 (6) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 6 (6) | 1 (1)
Somnolence (Nervous system disorders) | 7 (7) | 14 (14) | 14 (15) | 17 (18)
Dizziness (Nervous system disorders) | 9 (13) | 12 (16) | 14 (15) | 16 (17)
Headache (Nervous system disorders) | 14 (21) | 11 (14) | 6 (8) | 13 (16)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days